CLINICAL TRIAL: NCT07138690
Title: A Retrospective, Single-center Observational Study on Ultrasound-guided Centrally Inserted Central Catheters Catheter-related Bloodstream Infection and Catheters Failure in Adult Cardiac Surgical Patients.
Brief Title: Complications and Failure of Centrally Inserted Central Catheters in Cardiac Surgical Patients
Acronym: CICC-CS
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Raffaele Mandarano, Principal Investigator, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: CEAVC 26787
Record Dates: First submitted 2025-08-13; First posted 2025-08-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: CRBSI - Catheter Related Bloodstream Infection; Central Venous Catheter; Catheter Failure; Central Venous Catheter Complications
Keywords: catheter failure; CRBSI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac surgical patients: Cardiac surgical patients with ultrasound guided centrally inserted catheter into the internal jugular vein

SUMMARY:
Central venous catheters, or CVCs, are medical devices used to deliver medications and blood products directly into a patient's large veins. They are now an essential part of modern hospital care, but their use comes with potential complications.

Two of the most serious and well-studied complications are catheter-related bloodstream infections and catheter-related thrombosis (blood clots). These issues not only pose significant health risks to patients but also increase healthcare costs. Fortunately, the frequency of these complications has been reduced by following universally accepted prevention measures, such as:

Proper hand hygiene and skin disinfection before insertion

Using an ultrasound to guide the procedure

Applying best practices for ongoing catheter maintenance

Besides infections and blood clots, other complications like accidental displacement, lumen occlusion (blockage), or a suspected infection can lead to the early, or premature, removal of a CVC before the completion of the patient's treatment.

In patients undergoing cardiac surgery, CVCs are vital. They are used for general anesthesia, medication delivery, and continuous monitoring of a patient's heart and circulatory system. Because of this critical role, it's essential to constantly monitor the incidence of CVC-related complications in this patient population.

This single-center, retrospective study will investigate two primary objectives:

The frequency of catheter-related infections in adult patients undergoing cardiac surgery.

The frequency of premature catheter removals, or "catheter failures," in the same patient group.

The findings from this study will help improve the management of CVCs in cardiac surgery patients and reduce and prevent future complications.

DETAILED DESCRIPTION:
Over recent decades, numerous studies have examined the long-term complications associated with centrally inserted central catheters (CICCs). Among these, catheter-related bloodstream infections (CRBSIs) have been the most extensively investigated due to their association with increased mortality, prolonged hospital stays, and higher healthcare costs. More recently, premature catheter removal-commonly referred to as catheter failure-has emerged as a frequent yet underexplored complication of CICCs and other vascular access devices (VADs), given its contribution to increased patient risk and healthcare burden.

These findings have informed multiple national and international guidelines for CICC placement and management, resulting in significant advances in the prevention and management of CRBSIs and catheter-related thrombosis (CRT), the major causes of late catheter-related complications.

Currently, ultrasound-guided axillary venous access is considered the preferred central venous access site in intensive care units and, more broadly, in hospitalized patients to reduce CRBSI risk.

In cardiac surgical patients, a CICC is required for the administration of general anesthesia during surgery, as well as for intravenous infusions and medications during the postoperative stay in the intensive care unit and cardiac wards. Traditionally, the right internal jugular vein (IJV) has been favored-likely because it was the most accessible site for central venous cannulation in the pre-ultrasound era.

Current evidence shows that right IJV cannulation is associated with a lower risk of mechanical complications and thrombosis, whereas subclavian or axillary vein (SCV/AV) cannulation is linked to a reduced incidence of CRBSIs. However, SCV/AV access-particularly when performed via blind puncture-carries the risk of pinch-off syndrome and, in rare cases, catheter fracture due to compression between the clavicle and the first rib.

For these reasons, the right IJV remains the preferred site during cardiac surgery, while SCV/AV access may be favored postoperatively to lower infection risk and improve patient comfort.

Several factors specific to cardiac surgery further support the choice of the right IJV. These include the potential need for postoperative pacemaker implantation via the left subclavian vein, possible surgical interruption of the brachiocephalic vein during aortic procedures, the favorable anatomy of the right IJV for passage to the superior vena cava, and the elevated bleeding risk in patients requiring perioperative anticoagulation.

In cardiac surgery, the reported incidence of CRBSIs is 1-5%, comparable to that in ICU patients, while the incidence of catheter failure remains unknown. Given the persistent use of the right IJV in cardiac surgery-despite guidelines favoring axillary access-further research into outcomes associated with the IJV in this patient population is warranted.

A comprehensive investigation into the incidence and risk factors for CRBSIs and catheter failure in cardiac surgical patients is essential to optimize CICC management and improve patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years.
* Signed informed consent for contactable patients and those who will be attending the treatment center for follow-up visits.
* Patients undergoing elective or emergency cardiac surgery during the study period.
* Cardiac anesthesiologist performing the procedure with >2 years of experience in cardiac surgery and with >100 ultrasound-guided CICC placement procedures per year.
* Patient with a triple- or quad-lumen CICC placed in the right internal jugular vein.

Exclusion Criteria:

* Patients with active endocarditis.
* Patients with preoperative sepsis.
* Patients with infection confirmed by another source.
* Patients under 18 years of age.
* Patients who died within 7 days of surgery.
* Patients with a CICC already in place at the time of surgery.
* Cardiac anesthesiologist with less than 2 years of cardiac surgery experience and/or fewer than 100 procedures per year.
* Patients with a CICC placed in the left IJV, subclavian veins, or femoral veins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery performed at the study site with a ultrasound guided right internal jugular vein centrally inserted central catheter placed in the operating room.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
CRBSI | Perioperative
  Incidence of catheter related bloodstream infection. No of CRBSI/Total catheters*100. No of CRBSI/1000 catheter days.

SECONDARY OUTCOMES:
Catheter failure | Perioperative
  No of catheters removed (causes:CRBSI, CRT, suspected CRI, catheter malposition, catheter malfunction, accidental dislodgment, site competition)/Total catheters * 100

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Mandarano, MD, MSc, Principal Investigator — Azienda Ospedaliero-Universitaria Careggi
Locations (1):
- Cardiac ICU - Department of Anesthesia and Intensive Care - Careggi University Hospital, Florence, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Researchers, clinicians, or public health authorities conducting ethically approved studies aimed at improving patient care or health outcomes could request the data.

REFERENCES:
- [Background] Rockholt MM, Agrell T, Thorarinsdottir H, Kander T. Sustained low catheter related infection (CRI) incidence in an observational follow-up study of 9924 catheters using automated data scripts as quality assurance for central venous catheter (CVC) management. Infect Prev Pract. 2023 Feb 19;5(2):100273. doi: 10.1016/j.infpip.2023.100273. eCollection 2023 Jun. PMID 36926533
- [Background] Takashima M, Schults J, Mihala G, Corley A, Ullman A. Complication and Failures of Central Vascular Access Device in Adult Critical Care Settings. Crit Care Med. 2018 Dec;46(12):1998-2009. doi: 10.1097/CCM.0000000000003370. PMID 30095499
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Corley A, Royle RH, Marsh N, Larsen EN, Playford EG, McGrail MR, Runnegar N, Ware RS, Gavin NC, Alexandrou E, Murgo M, Gowardman JR, Regli A, Rickard CM. Incidence and risk factors for central venous access device failure in hospitalized adults: A multivariable analysis of 1892 catheters. J Hosp Med. 2024 Oct;19(10):905-917. doi: 10.1002/jhm.13414. Epub 2024 May 27. PMID 38800854
- [Background] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710
- [Background] Brescia F, Pittiruti M, Ostroff M, Spencer TR, Dawson RB. The SIC protocol: A seven-step strategy to minimize complications potentially related to the insertion of centrally inserted central catheters. J Vasc Access. 2023 Mar;24(2):185-190. doi: 10.1177/11297298211036002. Epub 2021 Jul 29. PMID 34320856
- [Background] Grant MC, Crisafi C, Alvarez A, Arora RC, Brindle ME, Chatterjee S, Ender J, Fletcher N, Gregory AJ, Gunaydin S, Jahangiri M, Ljungqvist O, Lobdell KW, Morton V, Reddy VS, Salenger R, Sander M, Zarbock A, Engelman DT. Perioperative Care in Cardiac Surgery: A Joint Consensus Statement by the Enhanced Recovery After Surgery (ERAS) Cardiac Society, ERAS International Society, and The Society of Thoracic Surgeons (STS). Ann Thorac Surg. 2024 Apr;117(4):669-689. doi: 10.1016/j.athoracsur.2023.12.006. Epub 2024 Jan 28. PMID 38284956
- [Background] Prachanpanich N, Morakul S, Kiatmongkolkul N. Effectiveness of securing central venous catheters with topical tissue adhesive in patients undergoing cardiac surgery: a randomized controlled pilot study. BMC Anesthesiol. 2021 Mar 8;21(1):70. doi: 10.1186/s12871-021-01282-0. PMID 33685394
- [Background] Greco G, Shi W, Michler RE, Meltzer DO, Ailawadi G, Hohmann SF, Thourani VH, Argenziano M, Alexander JH, Sankovic K, Gupta L, Blackstone EH, Acker MA, Russo MJ, Lee A, Burks SG, Gelijns AC, Bagiella E, Moskowitz AJ, Gardner TJ. Costs associated with health care-associated infections in cardiac surgery. J Am Coll Cardiol. 2015 Jan 6;65(1):15-23. doi: 10.1016/j.jacc.2014.09.079. PMID 25572505
- [Background] Vervoort D. Global cardiac surgery: a wake-up call. Eur J Cardiothorac Surg. 2019 May 1;55(5):1022-1023. doi: 10.1093/ejcts/ezy319. No abstract available. PMID 30260391
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee. Guidelines for the prevention of intravascular catheter-related infections. Am J Infect Control. 2011 May;39(4 Suppl 1):S1-34. doi: 10.1016/j.ajic.2011.01.003. No abstract available. PMID 21511081
- [Background] Mermel LA. Prevention of intravascular catheter-related infections. Ann Intern Med. 2000 Mar 7;132(5):391-402. doi: 10.7326/0003-4819-132-5-200003070-00009. PMID 10691590
- [Background] Tarricone R, Torbica A, Franzetti F, Rosenthal VD. Hospital costs of central line-associated bloodstream infections and cost-effectiveness of closed vs. open infusion containers. The case of Intensive Care Units in Italy. Cost Eff Resour Alloc. 2010 May 10;8:8. doi: 10.1186/1478-7547-8-8. PMID 20459753
- [Background] Raad II, Luna M, Khalil SA, Costerton JW, Lam C, Bodey GP. The relationship between the thrombotic and infectious complications of central venous catheters. JAMA. 1994 Apr 6;271(13):1014-6. PMID 8139059
- [Background] Pandit P, Sahni AK, Grover N, Dudhat V, Das NK, Biswas AK. Catheter-related blood stream infections: prevalence, risk factors and antimicrobial resistance pattern. Med J Armed Forces India. 2021 Jan;77(1):38-45. doi: 10.1016/j.mjafi.2019.07.002. Epub 2019 Oct 15. PMID 33487864
- [Background] Kalso E. A short history of central venous catheterization. Acta Anaesthesiol Scand Suppl. 1985;81:7-10. doi: 10.1111/j.1399-6576.1985.tb02313.x. PMID 3909712